CLINICAL TRIAL: NCT06708468
Title: Personalized Exercise Training for People With Rare Neuromuscular Disorders: a Multi-center, Evaluator-blinded, Two Arm, Randomized Controlled Study to Assess the Effects on Physical Function From Personalized Strength and Balance Exercise in a Rehabilitation Setting.
Brief Title: Personalized Training for People With Rare Neuromuscular Disorders
Acronym: PETRA-NMD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Universitetssykehuset i Nord-Norge HF (Unknown); Norwegian School of Sport Sciences (Other); Namsos Hospital (Other); Frambu Centre for Rare Disorders (Unknown); Vigør Rehabilitation Hospital (Unknown); Kastvollen Rehabilitation Centre (Unknown); Norwegian University of Science and Technology (Other); Haukeland University Hospital (Other); Molde Hospital (Other); Drammen sykehus (Other); Vikersund Bad Rehabiliteringssenter AS (Unknown); Røde Kors Haugland rehabilitation center (Other)
Responsible Party: Principal Investigator, Kristin Ørstavik, head of Section, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 760722
Record Dates: First submitted 2024-11-22; First posted 2024-11-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Neuromuscular Diseases (NMD); Charcot Marie Tooth Disease (CMT); Facioscapulohumeral Muscular Dystrophy; Myotonic Dystrophy Type 1 (DM1)
Keywords: personalized training; rehabilitation; rare-neuromuscular disorders; motor unit number estimation; neuromuscular ultrasound; dual-energy x-ray absorptiometry; activity tracking; metabolomics; dynamic balance
MeSH Terms: conditions — Neuromuscular Diseases; Charcot-Marie-Tooth Disease; Muscular Dystrophy, Facioscapulohumeral; Myotonic Dystrophy | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a multi-site randomized control trial with two study arms - interventional and control group that will be investigated pre-and-post four-month intervention, and at 10-month and 16-month for follow-up. The participants will involve three different rare-NMDs (CMT, FSHD, DM1) from the four health regions of Norway - South-Eastern, Northern, Central, and Western. The participants will be randomly allocated to either the intervention or control group. The interventional group will undergo a personalized four month exercise training program at a rehabilitation centre followed by at-home digital exercises; whereas, the control group will receive usual care. The two groups will be stratified by study site, diagnosis and sex.
Who Masked: Outcomes Assessor
Masking Description: The evaluators will be blinded to the treatment group of the participants. It is not possible to blind the participants themselves; however, they will be asked not to share their group allocation with the others, including the evaluators. A staff member may unblind the intervention assignment for any participant with a serious adverse event.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The experimental group receives four-months of exercise-based intervention
  Interventions: Other: Exercise
- Control (Active Comparator): The control group follows usual care
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Exercise — The intervention includes 12-day personalized exercise program set in a rehabilitation center, followed by a three-month digital intervention and then a second 12-day personalized exercise program in a rehabilitation center.
  Other Names: Personalized Exercise
  Arms: Intervention
Other: Usual Care — Usual care includes appointments at hospitals and in the community health system according to what has been recommended to that individual
  Arms: Control

SUMMARY:
The goal of this study is to investigate the effects of personalized exercise treatment on dynamic balance and physical function in comparison with regular follow-up in adults with rare-neuromuscular disorders: Charcot-Marie-Tooth (CMT), Facioscapulohumeral Muscular Dystrophy (FSHD), and Myotonic Dystrophy Type 1 (DM1).

The key objectives are:

1. To investigate if the intervention group experiences improvements in dynamic balance that are superior to the control group
2. To investigate if the intervention group experiences long-term improvements in dynamic balance that are superior to the control group during the follow-up
3. To investigate if improvements in dynamic balance are associated with improvements in physical activity, body composition, estimated motor units, metabolomics, muscle echnogenecity and volume, and other indicators of health and quality of life.

This is a national study and will involve 120 individuals with rare-neuromuscular disorders from Norway's four health regions.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of either FSHD, DM1 or CMT
* 18-70 years of age at the time of signing the informed consent.
* Any gender
* Ability to stand, rise from a chair and walk at least 10 meters with or without any need of assistive devices
* Indication for rehabilitation as confirmed by the treating neurologist or physiotherapist
* Ability to understand and follow instructions in Norwegian
* Capable of giving signed informed consent

Exclusion Criteria:

* Pregnancy or planning to become pregnant
* Any other neurological or non-neurological disorders affecting physical capacity, such as disabling arthritis, severe heart-failure/cardiomyopathy, on-going cancer treatment
* Alcohol or drug abuse as per their medical chart
* History of non-compliance to medical advice/follow-up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Dynamic balance assessed using Mini-Balance Evalulation Systems Test (Mini-BESTest) | Baseline, 4-month (primary), follow-up at 10-month and 16-month (only interventiongroup)
  The primary outcome measure will be change in dynamic balance from pre-intervention to post-intervention. In addition, there will be two follow-up assessments.

SECONDARY OUTCOMES:
Fatigue severity scale | Baseline, 4-month, 10-month and 16-month (only intervention-group)
  Measurements of fatigue, 9 questions on a scale from 1 to 7. And a visual analogue fatigue scale
Clinical measures of strength and function | Baseline 4-month, 10-month and 16-month (only intervention group)
  manual muscle testing, 30-s sit-to-stand, functional strength of neck and trunk, arm and hand function (9-HPT, Box and Block), walking function (10-mWT and 100-mTT), grip and pinch strength using dynamometers.
Global Metabolomics | Baseline, 4-month, 10-month
  dried blood samples for extracting signal metabolites of known importance in characterizing the metabolic status (e.g. lactate, amino acids, and fatty acids)
Dual Energy X-ray Absorptiometry | 4-month, 10-month and 16-month
  body composition from different regions of the body
Neuromuscular ultrasound | 4-month, 10-month and 16-month
  Ultrasound imaging of selected muscles in the trunk, upper- and lower extremities scored using visual and/or quantitative grey-scale echogenicity analysis tools. Only collected in participants with FSHD and DM1.
Physical activity | 4-month, 10-month and 16-month
  tri-axial AX3 accelerometers, and monitoring pain, and activity and sleep diaries. Only collected in participants from Helse Sør-Øst.
Motor unit number estimation | Baseline 4-month, 10-month and 16-month (only intervention-group)
  Estimating the number of motor units using non-invasive peripheral nerve stimulation and surface electromyography recordings. Only for participants with CMT at Helse Sør-Øst.
ABC-scale | Basleine, 4 month, 10 month, 16 month (only intervention group)
  Activities- specific balance confidence scale.
PROMIS-29 | Baseline, 4 month, 10 month and 16 month (only intervention group)
  Questionnaire with 7 domains and a numeric rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Ørstavik, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (5):
- Norway (5):
  - Haukeland University Hospital, Bergen
  - Helse Møre and Romsdal HF (Molde Hospital), Molde
  - Namsos Hospital, Namsos
  - Oslo University Hospital, Oslo
  - University Hospital of North Norway, Tromsø

IPD SHARING:
Plan to Share IPD: Undecided